CLINICAL TRIAL: NCT00147953
Title: A Phase II Study of Rituximab Plus Low-Dose Radiotherapy in Patients With Relapsed Non-Hodgkin's Lymphoma
Brief Title: Study to Evaluate the Efficacy of Rituximab in Combination With Low-dose Radiotherapy in Patients With Relapsed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ritux plus TNI
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NHL; Lymphoma; Radiotherapy; Rituximab; Palliative treatment
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab
Procedure: Total nodal irradiation

SUMMARY:
This study aims to assess the short term efficacy of a combination of rituximab and low-dose radiotherapy in patients with non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Rituximab and low-dose total-nodal irradiation both have shown promising activity in patients with NHL. Moreover, the radiolabelled antibody Zevalin has been approved for the treatment of relapsed NHL. The patients in this study have a poor prognosis. The treatment strategy aims to control the disease and to ameliorate disease related symptoms with minimal toxicity. Both, rituximab and low-dose radiotherapy are associated with minor toxicity if applied alone.

The primary objective of the study is therefore to assess the short term efficacy of a combination of rituximab and low-dose radiotherapy in patients with non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* B-cell non-Hodgkin's lymphoma
* At least one prior antitumor therapy
* ECOG performance status 0-2
* No major organ dysfunction
* Written informed consent

Exclusion Criteria:

* The following histologies are excluded: Burkitt's lymphoma, mantle-cell lymphoma, primary CNS-lymphoma, HIV-associated lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Overall response rate (complete and partial response rate)

SECONDARY OUTCOMES:
Toxicity
Time to progression
Response duration
Quality-of-Life

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Principal Investigator — University of Cologne; R.-P. Mueller, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, North Rhine-Westphalia, Germany